CLINICAL TRIAL: NCT04901897
Title: A Study to Evaluate the Product Performance of a New Silicone Hydrogel Contact Lens
Brief Title: Product Performance of a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 893
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- kalifilcon A (Experimental): kalifilcon A daily disposable contact lens
  Interventions: Device: kalifilcon A
- delefilcon A (Active Comparator): DAILIES TOTAL1® (delefilcon A) daily disposable contact lenses
  Interventions: Device: delefilcon A
- senofilcon A (Active Comparator): Acuvue Oasys® 1-Day with HydraLuxe™ (senofilcon A) daily disposable contact lens
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: kalifilcon A — kalifilcon A daily disposable contact lens
  Arms: kalifilcon A
Device: delefilcon A — DAILIES TOTAL1® (delefilcon A) daily disposable contact lenses
  Arms: delefilcon A
Device: senofilcon A — Acuvue Oasys® 1-Day with HydraLuxe™ (senofilcon A) daily disposable contact lens
  Arms: senofilcon A

SUMMARY:
The objective of this study is to evaluate the product performance of kalifilcon A, compared to the Johnson & Johnson Acuvue Oasys® 1-Day with HydraLuxe™ (senofilcon A) daily disposable contact lens and Alcon DAILIES TOTAL1® (delefilcon A) daily disposable contact lenses when worn by current soft contact lens wearers on a daily disposable wear basis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old on the date the ICF is signed and have capacity to provide voluntary informed consent.
* myopic and require lens correction from -0.50 to -6.00 Diopter (D) with 0.25 D steps, in each eye.
* correctable through spherocylindrical refraction and with soft spherical contact lenses to 32 letters (0.3 logarithm of the minimum angle of resolution [logMAR]) or better (2 meters distance, high-contrast chart) in each eye.
* free of any anterior segment disorders.
* adapted soft contact lens wearers and willing to wear their study lenses for at least 8 hours per day on a daily disposable wear basis for approximately 2 weeks.
* access to internet connection and personal email to send/receive emails.
* habitually wear either Alcon's Air Optix Aqua, Air Optix with HydraGlyde, Air Optix Night & Day, Bausch + Lomb's PureVision 2, Bausch + Lomb ULTRA, CooperVision's Biofinity, Johnson & Johnson Acuvue Oasys® with HydraClear™, or Acuvue Vita soft contact lenses.

Exclusion Criteria:

* participating in any drug or device clinical investigation within 2 weeks prior to entry into this study (Screening/Dispensing Visit) and/or during the period of study participation.
* have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* have any systemic or ocular disease currently affecting ocular health in the Investigator's opinion may have an effect on ocular health during the course of the study.
* using any systemic, topical or topical ocular medications that will in the Investigator's opinion, affect ocular physiology or lens performance.currently wear daily disposable, monovision, multifocal, or toric contact lenses.
* refractive astigmatism of greater than 0.75 D in either eye.
* anisometropia (spherical equivalent) of greater than 2.00 D.
* amblyopic.
* have had any corneal surgery (e.g., refractive surgery).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 805 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, Study Director — Bausch & Lomb Incorporated
Locations (35):
- United States (35):
  - Bausch Site 433, Birmingham, Alabama
  - Bausch Site 431, Scottsdale, Arizona
  - Bausch Site 406, Azusa, California
  - Bausch Site 430, Los Angeles, California
  - Bausch Site 419, San Diego, California
  - Bausch Site 435, San Francisco, California
  - Bausch Site 432, Sunnyvale, California
  - Bausch Site 409, Torrance, California
  - Bausch Site 416, Denver, Colorado
  - Bausch Site 415, Jacksonville, Florida
  - Bausch Site 434, Jacksonville, Florida
  - Bausch Site 405, Sarasota, Florida
  - Bausch Site 412, Decatur, Georgia
  - Bausch Site 437, Honolulu, Hawaii
  - Bausch Site 401, ‘Aiea, Hawaii
  - Bausch Site 414, Leavenworth, Kansas
  - Bausch Site 413, Portland, Maine
  - Bausch Site 421, Sterling Heights, Michigan
  - Bausch Site 429, Edina, Minnesota
  - Bausch Site 422, Raytown, Missouri
  - Bausch Site 407, St Louis, Missouri
  - Bausch Site 418, Warrensburg, Missouri
  - Bausch Site 424, Jamestown, New York
  - Bausch Site 403, Vestal, New York
  - Bausch Site 417, Raleigh, North Carolina
  - Bausch Site 411, Fargo, North Dakota
  - Bausch Site 423, Miamisburg, Ohio
  - Bausch Site 425, West Chester, Ohio
  - Bausch Site 428, Grants Pass, Oregon
  - Bausch Site 420, State College, Pennsylvania
  - Bausch Site 427, Warwick, Rhode Island
  - Bausch 410, Brentwood, Tennessee
  - Bausch Site 408, Memphis, Tennessee
  - Bausch Site 404, Nashville, Tennessee
  - Bausch Site 426, League City, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kalifilcon A | Delefilcon A | Senofilcon A
Started | 398 | 202 | 205
Completed | 393 | 200 | 203
Not Completed | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kalifilcon A | Delefilcon A | Senofilcon A | Total
Number analyzed (Participants) | 398 | 202 | 205 | 805
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (5.72) | 30.0 (6.11) | 29.3 (5.78) | 30.3 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 125 | 140 | 527
  Male | 136 | 77 | 65 | 278
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 56 | 30 | 26 | 112
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 1 | 8
  Black or African American | 47 | 17 | 25 | 89
  White | 281 | 147 | 146 | 574
  More than one race | 10 | 3 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in logMAR Contact Lens Visual Acuity
Description: logMAR is the logarithm of the minim angle of resolution
Time Frame: Baseline, 2 Week Follow up
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Kalifilcon A | Delefilcon A | Senofilcon A
Number analyzed (Participants) | 398 | 202 | 205
Number analyzed (eyes) | 796 | 404 | 410
logMAR | -0.056 (0.0727) | -0.069 (0.0733) | -0.069 (0.0718)

2. Primary Outcome: Percentage of Participants in the Test Lens Group Agreeing With the Statement "Are Comfortable Throughout the Day"
Time Frame: 2 Week Follow up
Population: Participants with 2 week follow up and responded to the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Kalifilcon A | Delefilcon A | Senofilcon A
Number analyzed (Participants) | 391 | 200 | 199
Participants | 317 | 160 | 166

3. Primary Outcome: Percentage of Participants in the Test Lens Group Agreeing With the Statement "Provide Clear Vision Throughout the Day"
Time Frame: 2 Week Follow up
Population: Participants with 2 week follow up and responded to the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Kalifilcon A | Delefilcon A | Senofilcon A
Number analyzed (Participants) | 392 | 201 | 201
Participants | 358 | 184 | 188

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events occurring after signing of informed consent and through the participant's end of participation in the study were reported.
Arm/Group | Kalifilcon A | Delefilcon A | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/398 | 0/202 | 0/205
Serious Adverse Events (participants affected / at risk) | 0/398 | 0/202 | 0/205
Other Adverse Events (participants affected / at risk) | 0/398 | 0/202 | 0/205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04901897/Prot_SAP_000.pdf